CLINICAL TRIAL: NCT01002235
Title: A Phase I/II, Open Label, Dose-Escalation Study to Assess the Safety and Tolerability of Engensis (VM202) in Patients With Painful Diabetic Peripheral Neuropathy
Brief Title: Gene Therapy for Painful Diabetic Neuropathy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Helixmith Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VMDN-001/G
Record Dates: First submitted 2009-10-24; First posted 2009-10-27 (Estimated); Results first posted 2025-06-15 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-08

CONDITIONS: Painful Diabetic Peripheral Neuropathy
Keywords: Diabetic; Neuropathy; Peripheral; diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Dose Ranging
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1 (Experimental): Two divided doses of VM202 injected into the calf muscle on Day 0 and Day 14 for a total dose of 4 mg.
  Interventions: Biological: VM202
- Cohort 2 (Experimental): Two divided doses of VM202 injected into the calf muscle on Day 0 and Day 14 for a total dose of 8mg.
  Interventions: Biological: VM202
- Cohort 3 (Experimental): Two divided doses of VM202 injected into the calf muscle on Day 0 and Day 14 for a total dose of 16mg.
  Interventions: Biological: VM202

INTERVENTIONS:
Biological: VM202 — Intramuscular injections in the calf on Day 0 and Day 14.

SUMMARY:
The purpose of this open label, Phase I/II, dose-escalation, 3-cohort, multicenter, 12-month study, is to assess the safety and tolerability of injecting Engensis (VM202) in the leg muscle in patients with painful diabetic peripheral neuropathy (DPN). The study will also assess the potential of VM202 to reduce the pain associated with diabetic peripheral neuropathy.

DETAILED DESCRIPTION:
Peripheral neuropathy is a serious complication of diabetes. This form of neuropathy carries a high risk of pain, trophic changes and autonomic dysfunction.

Currently, there are no approved drugs or interventional strategies known to halt or reverse the progression of painful diabetic peripheral neuropathy (DPN). Treatments target pain reduction, physical function improvement, reduction of psychological distress, and quality of life improvements.

There is currently no effective treatment for diabetic neuropathy, and good glycemic control is the only way to minimize the risk of occurrence. Clearly, it would be desirable to prevent, impede, or reverse the disrupting and often life-threatening manifestations of peripheral neuropathy by stimulating growth or regeneration of peripheral nerve axons.

The purpose of this open label, dose-escalation, 3-cohort study is to assess the safety and tolerability of injecting Engensis (VM202) in the leg muscle in patients with painful diabetic peripheral neuropathy. The study will also assess the potential of VM202 to reduce the pain associated with diabetic peripheral neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years to 75 years
* Documented history of Type I or II diabetes with current treatment control (glycosylated hemoglobin A1c of ≤ 10.0%)
* Diagnosis of painful diabetic peripheral neuropathy in both lower extremities
* The physical examination component of the Michigan Neuropathy Screening Instrument Score (MNSI) is ≥ 3 at Screening
* Visual analog scale (VAS) score of ≥ 4 cm at Screening (0 cm = no pain - 10 cm worst imaginable pain)
* Stable treatment of diabetes for at least 3 months with no anticipated changes in medication regimen, and no new symptoms associated with diabetes
* Lower extremity pain for at least 6 months
* If female of childbearing potential, negative pregnancy test at screening and using acceptable method of birth control during the study.

Exclusion Criteria:

* Peripheral neuropathy caused by condition other than diabetes;
* Other pain more severe than neuropathic pain;
* Progressive or degenerative neurological disorder;
* Myopathy;
* Inflammatory disorder of the blood vessels (inflammatory angiopathy, such as Buerger's disease);
* Active infection;
* Chronic inflammatory disease (e.g. Crohn's, Rheumatoid Arthritis)
* Positive HIV or HTLV at Screening
* Positive Hepatitis B or C as determined by Hepatitis B core antibody (HBcAB), antibody to Hepatitis B antigen (IgG and IgM; HbsAB), Hepatitis B surface antigen (HBsAg) and Hepatitis C antibodies (Anti-HCV), at Screening or known immunosuppression or on chronic treatment with immunosuppressive drugs, chemotherapy or radiation therapy
* Stroke or myocardial infarction within last 6 months;
* Ophthalmologic conditions pertinent to proliferative retinopathy or conditions that preclude standard ophthalmologic examination:

  * Cataract surgery within 6 months of trial;
  * Vascular lesions of the anterior segment of the eye (infection or ulceration of the cornea, rubeotic glaucoma, etc);
  * Vascular lesions of the posterior segment of the eye or proliferative retinopathy, macular edema, s/p photocoagulation for macular edema or proliferative retinopathy; sickle cell retinopathy, ischemic retinopathy due to retinal venous stasis or carotid artery disease;
  * Choroidal angiogenesis; and
  * Large elevated choroidal nevi, choroidal vascular tumors (choroidal hemangioma), or melanomas.
* Specific laboratory values at Screening including: Hemoglobin < 9.0 g/dL, WBC < 3,000 cells per microliter, platelet count <75,000/mm3, Creatinine > 2.0 mg/dL; GFR < 50, AST and/or ALT > 2 times the upper limit of normal or any other clinically significant lab abnormality which in the opinion of the investigator should be exclusionary;
* Use of gamma-linolenic acid (GLA), alpha lipoic acid or any other high dose dietary antioxidant supplement for symptomatic relief of DPN;
* Uncontrolled hypertension as defined as sustained systolic blood pressure (SBP) > 200 mmHg or diastolic BP (DBP) > 110 mmHg at baseline/screening evaluation;
* Patients with history of or new screening finding of malignant neoplasm except basal cell carcinoma or squamous cell carcinoma of the skin (if excised and no evidence of recurrence);
* Malignant tumors or abnormal screening test suspicious for cancer, or patients in whom screening exams indicate possible occult malignancy unless malignancy has been ruled out. Patients with family history of colon cancer in any first degree relative unless they have undergone a colonoscopy in the last 12 months with negative findings;
* Elevated PSA unless prostate cancer has been excluded;
* Subjects requiring > 81 mg daily of acetylsalicylic acid; If > 81 mg are taken at screening, subjects may be enrolled if willing/able to switch to another medication;
* Major psychiatric disorder in past 6 months;
* History of drug or alcohol abuse / dependence in the past 2 years;
* History of recent tobacco abuse (within past 5 years);
* BMI > 38 kg/m2;
* Use of an investigational drug or treatment in past 12 months; and
* Unable or unwilling to give informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-02; Primary Completion 2011-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Kessler, M.D., Principal Investigator — Northwestern Memorial Hospital
Locations (2):
- United States (2):
  - Diablo Clinical Research Hospital, Walnut Creek, California
  - Northwestern Memorial Hospital, Chicago, Illinois

REFERENCES:
- [Background] Ajroud-Driss S, Christiansen M, Allen JA, Kessler JA. Phase 1/2 open-label dose-escalation study of plasmid DNA expressing two isoforms of hepatocyte growth factor in patients with painful diabetic peripheral neuropathy. Mol Ther. 2013 Jun;21(6):1279-86. doi: 10.1038/mt.2013.69. Epub 2013 Apr 23. PMID 23609019

RESULTS

PARTICIPANT FLOW:
Groups:
- Engensis 4 mg: Subjects received Intramuscular injections of Engensis to the calf on Days 0 and 14
- Engensis 8 mg: Subjects received Intramuscular injections to the calf on Days 0 and 14
- Engensis 16 mg: Subjects received Intramuscular injections of Engensis on Days 0 and 14
Period: Overall Study
Arm/Group | Engensis 4 mg | Engensis 8 mg | Engensis 16 mg
Started | 4 | 4 | 4
Completed | 4 | 4 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population including any subject who received all assigned dose of Engensis and had evaluable data at a follow-up visit
Groups:
- Total: Total of all reporting groups
Arm/Group | Engensis 4 mg | Engensis 8 mg | Engensis 16 mg | Total
Number analyzed (Participants) | 4 | 4 | 4 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (7.0) | 61.3 (7.1) | 54.8 (12.4) | 58.8 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 4 | 4 | 4 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 4 | 3 | 4 | 11
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Treatment-emergent Adverse Events for Participants Who Received Engensis 4 mg, 8 mg, or 16 mg
Description: Treatment-emergent adverse events are any adverse events that occurred after the first dose of Engensis (VM202).
  This is a dose escalation study. Cohorts of increasing dose will be enrolled sequentially. Dose escalation decisions (permission to treat at higher doses) will be made by the Data Safety Monitoring Board based on review of adverse events and on the occurrence of dose limiting toxicities in each cohort. The decision to proceed to the next higher dose cohort will be made according to the scheme described in the protocol.
Time Frame: Day 0 to Day 365
Population: The Safety Population included all participants who received at least one dose of Engensis (VM202) from Day 0 to Day 365
Measure: Count of Participants; unit: Participants
Groups:
- Engensis 4 mg; Engensis 8 mg: Subjects received Intramuscular injections of Engensis (VM202) to the calf on Days 0 and 14
- Engensis 16 mg: Subjects received Intramuscular injections of Engensis (VM202) on Days 0 and 14
Arm/Group | Engensis 4 mg | Engensis 8 mg | Engensis 16 mg
Number analyzed (Participants) | 4 | 4 | 4
Participants
  Subjects with any TEAEs | 3 | 2 | 2
  Back pain | 1 | 1 | 0
  Musculoskeletal pain | 0 | 0 | 1
  Dry eye | 1 | 0 | 0
  Retinal vascular disorder | 0 | 0 | 1
  Diarrhoea | 1 | 0 | 0
  Dry mouth | 1 | 0 | 0
  Dyspepsia | 1 | 0 | 0
  Sinusitis | 0 | 1 | 0
  Viral infection | 0 | 0 | 1
  Injection site reaction | 1 | 0 | 0
  Foot fracture | 0 | 0 | 1
  Benign prostatic hyperplasia | 0 | 1 | 0
  Ingrowing nail | 1 | 0 | 0

2. Secondary Outcome: Percent Change From Baseline in Visual Analog Scale Pain Scores
Description: Percent change in median Visual Analog Scale Pain Scores from baseline (Day 0). The Visual Analog Scale Pain scoring instrument is a 10-cm line, oriented horizontally, with the left end (0 cm, is 0 Percent) indicating "no pain" and the right end (10 cm, is 100 percent) representing "pain as bad as it can be".
  The Change from Baseline of the Visual Analog Scale Pain Score is the difference between the Day 0 and the Days 90, 180 and 365 scores.
  A negative difference in the Change from Baseline of the Visual Analog Scale Pain Scores, indicates an improvement (reduction of pain severity) of the treated groups Visual Analog Score.
Time Frame: Days 0, 90, 180, and 365
Population: Change from Baseline (Day 0) to visits Day 90, Day 180, and Day 365, in the Intent-to-treat (ITT) population participants who received all assigned doses of Engensis and had evaluable data at a follow-up visit
Measure: Median (Standard Deviation); unit: percentage of Change from Baseline
Arm/Group | Engensis 4 mg | Engensis 8 mg | Engensis 16 mg
Number analyzed (Participants) | 4 | 4 | 4
percentage of Change from Baseline
  Day 90 | -19.19 (71.53) | -40.76 (28.55) | -40.15 (21.50)
  Day 180 | -26.16 (84.35) | -58.40 (39.36) | -57.07 (30.26)
  Day 365 | -42.27 (108.26) | -67.57 (47.56) | -46.97 (29.01)

ADVERSE EVENTS:
Time Frame: 365 days
Arm/Group | Engensis 4 mg | Engensis 8 mg | Engensis 16 mg
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 3/4 | 2/4 | 2/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Engensis 4 mg (N=4) | Engensis 8 mg (N=4) | Engensis 16 mg (N=4)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 1 (2) | 0 (0) | 0 (0)
Retinal vascular disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Injection site reaction (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2010-09-23): https://cdn.clinicaltrials.gov/large-docs/35/NCT01002235/Prot_SAP_ICF_000.pdf